CLINICAL TRIAL: NCT04981002
Title: Analysis of the Accuracy of Telemedicine-guided Orthopedic Self-examination Compared to Face-to-face Assessment in an Emergency Care Unit: a Randomized Study
Brief Title: Telemedicine and Face-to-face Consultations Diagnostic Accuracy Comparison in Orthopedic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 46603821.9.0000.0071
Record Dates: First submitted 2021-07-21; First posted 2021-07-28 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2021-07

CONDITIONS: Orthopedic Patients
Keywords: Telemedicine; Orthopedics; Trauma; Emergency Room
MeSH Terms: conditions — Wounds and Injuries; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult patients with orthopedic complaints - telemedicine self exam before face-to-face evaluation (Active Comparator): First care will be performed via telemedicine with a clinical physician, guiding self-examination guided by telemedicine. After the remote consultation, a face-to-face evaluation will be performed with an orthopedist, according to institutional protocol.
  Interventions: Other: Telemedicine Consultation with self orthopedic exam; Other: Face-to-face Consultation
- Adult patients with orthopedic complaints - only face-to-face evaluation (Active Comparator): Face-to-face care with an orthopedist, according to institutional protocol.
  Interventions: Other: Face-to-face Consultation

INTERVENTIONS:
Other: Telemedicine Consultation with self orthopedic exam — Brief telemedicine consultation, with self orthopedic exam,blinded to subsequent face-to-face evaluation.
  Arms: Adult patients with orthopedic complaints - telemedicine self exam before face-to-face evaluation
Other: Face-to-face Consultation — Direct face-to-face evaluation (without telemedicine consultation before).

SUMMARY:
Adult patients with acute complaints related to the musculoskeletal system are prevalent and correspond to a large percentage of visits to Emergency Care Units (UPA), often performed by general practitioners. These patients, in most cases, present complaints associated with low-complexity trauma, which can be diagnosed through targeted physical examination and treated with basic guidelines (behavioral/medicinal). The diagnosis of a more complex fracture or injury requires an assessment by an orthopedist. Currently, patients with orthopedic complaints are often seen by telemedicine, but there are no studies that have compared the diagnostic accuracy of remote assessment with standard face-to-face assessment. Telemedicine is a recognized medical care strategy used for various situations, including as a virtual emergency service. Despite the current widespread use, there are few studies that have evaluated the diagnostic accuracy of telemedicine compared to face-to-face evaluation, and there are no specific studies in patients with orthopedic symptoms. Scientific evidence of high diagnostic accuracy in telemedicine care can support the investment and expansion of this modality, expanding and facilitating the access of patients to the health service, with a reduction in costs and the rational use of resources. The objective of the study is to analyze the diagnostic accuracy of telemedicine-guided self-examination compared to a face-to-face medical evaluation at the UPA in adult patients with orthopedic complaints. Secondary objectives are: evaluation of medical care time, indication of additional tests, guidance, medical prescription, proposed destination after completion of care, cost and patient satisfaction. It is a a randomized, prospective, single-center study carried out in the telemedicine and UPA sectors of Hospital Israelita Albert Einstein. Randomization will be 1:1 and patients will be allocated in the Tele group (evaluation by telemedicine followed by face-to-face evaluation) or in the Standard group (in-person evaluation). The sample calculated for non-inferiority was 50 patients in each group.

DETAILED DESCRIPTION:
Randomized, prospective, single-center study carried out in the telemedicine sectors and emergency care unit of Hospital Israelita Albert Einstein, Ibirapuera Unit. The randomization will be 1:1, from the commercial application Randomizer ®, by the member of the project Renata Vidigal Correia.

After randomization, patients will be included in one of two possible groups:

1. TELE Group: first care will be provided via telemedicine with a clinical physician, guiding self-examination guided by telemedicine. After the remote consultation, a face-to-face evaluation will be carried out with an orthopedist, according to institutional protocol.
2. GrupoSTANDARD: Face-to-face care with an orthopedist, according to institutional protocol.

The face-to-face evaluation will be carried out by the local UPA medical and orthopedic care team and the telemedicine evaluation by the fixed medical team of the HIAE service responsible for urgency/emergency care.

The study will be of non-inferiority with evaluation of accuracy in both groups, since the telemedicine group, after completion of care, will pass the face-to-face consultation (gold standard).

Both in face-to-face and telemedicine assessments, clinical data, final diagnosis, destination, total time of care, guidance, complementary exams and prescription will be computed. In the face-to-face evaluation, additional exams and medications received in situ will also be computed. The final diagnoses will receive nomenclature according to the International Statistical Classification of Diseases and Related Health Problems - ICD 10 (requirement of institutional records - Cerner) and will be grouped according to the equivalence of the syndromic diagnosis. The diagnosis of the face-to-face evaluation is made following institutional protocols based on extensive medical literature and approved by the institutional clinical staff, being representative of current medical practice and will be considered the gold standard diagnosis.

The total service time in minutes will be evaluated, verifying if telemedicine can change the total medical service time. The fee for complementary exams will be counted in the number of exams requested and their categorization (laboratory exam or imaging exam); the quantification in number and its categorization (behavioral measures, cryotherapy guidelines and new medical evaluation if necessary) of the guidelines; categorization of prescription (only symptomatic or medication in the UPA); destination categorization (high - item valid for both services, hospitalization - valid item for face-to-face care, search for the ER - valid item for telemedicine care), hospital cost (measured by the need for immobilization/complementary tests), and indication of additional tests .

The final diagnosis will be considered by the official report of the radiologist based on the imaging exams performed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Patient with orthopedic complaints according to the above diagnostic criteria, by the triage nurse.
* Signing the informed consent form.

Exclusion Criteria:

* Return to the UPA for maintenance or aggravation of the complaint;
* Age > 65 years;
* Patient with emergency room criteria by the evaluation of the triage nursing.
* Postoperative period of orthopedic surgery < 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of telemedicine diagnosis in adult patients with orthopedic complaints | through study completion, an average of 1 year
  The patient will be evaluated by telemedicine and / or face-to-face consultation and at the end will receive the diagnosis, which will be assigned the ICD code for orthopedic complaints. At the end, these ICDs will be grouped by the same clinical significance (M54: Neck pain and Low back pain; T11-T13: Extremity contusion; S93: Ankle Sprain) and will be compared between the two consultation methods (telemedicine versus face-to-face consultation).

SECONDARY OUTCOMES:
Time of medical care | through study completion, an average of 1 year
  Comparison of time (minutes) of medical care between telemedicine and face-to-face consultation.
Rate of indication for complementary exams | through study completion, an average of 1 year
  Comparison of rate (percentage) of indication for complementary exams between telemedicine and face-to-face consultation.
Types of requested exams | through study completion, an average of 1 year
  Comparison of types of requested exams (percentage) between telemedicine and face-to-face consultation.
Medical prescription | through study completion, an average of 1 year
  Comparison of medical prescription after completion of the service between telemedicine and face-to-face consultation.
Proposed destination after completion of the service | through study completion, an average of 1 year
  Comparison of proposed destination (percentage of discharge or hospitalization) after completion of the service between telemedicine and face-to-face consultation.
Total hospital cost after completion of care | through study completion, an average of 1 year
  Comparison of total hospital cost after completion of care (Real and Dollar) between telemedicine and face-to-face consultation.
Patient satisfaction | through study completion, an average of 1 year
  Comparison of patient satisfaction (percentage) between telemedicine and face-to-face consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Noel HS Oizerovici Foni, MD, Principal Investigator — Telemedicine Department, Hospital Israelita Albert Einstein, Sao Paulo, Brazil
Locations (1):
- Hospital Israelita Abert Einstein, São Paulo, Brazil

REFERENCES:
- [Derived] Foni NO, Accorsi TAD, Correia RFV, Moreira FT, Lima KA, Morbeck RA, Souza JL Jr, Pedrotti CHS, Wolosker N; TeleORTHOPEDICS Trial. Guideline-Based Telemedicine Assessment of Orthopedic Low-Risk Conditions by General Practitioners is Not Inferior to that of Face-to-Face Consultations with Specialists in the Emergency Department: A Randomized Trial. Telemed J E Health. 2024 Dec;30(12):2859-2869. doi: 10.1089/tmj.2024.0312. Epub 2024 Aug 21. PMID 39166332